CLINICAL TRIAL: NCT06321705
Title: Expanded Access, Open-Label, Safety Extension Study for Patients That Have Completed Parent Study CS1-003 and Who Are Judged by the Investigator to Benefit From Continued CS1 Treatment
Brief Title: Safety and Efficacy of Continued CS1 Treatment of Patients With Pulmonary Arterial Hypertension
Status: Available | Type: Expanded Access
Sponsor: Cereno Scientific AB (Industry)
Collaborators: Worldwide Clinical Trials (Other); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: CS1-004
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; CardioMEMS
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: CS1 — CS1 delayed release capsules will be supplied with 160 mg active pharmaceutical ingredient (API) per capsule. Three dose levels will be administered in this expanded access study at the same dose the patient received in the parent study (CS1-003) of 480 mg, 960 mg, or 1920 mg. All patients will later have the option to be titrated to the most efficacious and safe dose determined from the ongoing CS1-003 study when completed.

SUMMARY:
CS1-004 will be an extension of the CS1-003 Study. The primary objective of the CS1-004 study is to evaluate long-term safety and tolerability of continued treatment with CS1.

DETAILED DESCRIPTION:
CS1-004 will be an extension of the CS1-003 Study. The primary objective of the CS1-004 study is to evaluate long-term safety and tolerability of continued treatment with CS1. The exploratory objectives are to evaluate clinical benefit by using Cardio-Microelectromechanical system (CardioMEMS), echocardiography, cardiac magnetic resonance imaging, right heart catheterization, quality of life assessments, and actigraphy to measure changes in clinical response with continued treatment with CS1 in patients with Pulmonary Arterial Hypertension (PAH).

Up to 30 patients are planned for enrollment in the ongoing phase 2 Study CS1-003; thus up to 30 patients could participate in Study CS1-004, if they completed the parent study, tolerated CS1 treatment, and in the investigator's judgement the benefits of continued treatment with CS1 outweigh the risk. Note that as the parent study is ongoing; thus, some patients will directly roll- over into Study CS1-004 with no disruption in CS1 treatment, while other patients that have already completed Study CS1-003, will need to be restarted on CS1. On a yearly basis, the principal investigator will determine if a patient continues the expanded access study for a subsequent year based on safety, tolerability, and clinical benefit of CS1. Continuation of the expanded access study will also be evaluated on a yearly basis by Cereno Scientific (Sponsor).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has derived benefit from CS1 treatment in parent Study CS1-003 based on the Investigator's judgement and the benefit of continued CS1 treatment outweighs the risk or the patient could benefit from continued treatment with CS1.
2. Patient must be willing and able to sign a written informed consent prior to any study-related procedures and able to understand and follow instructions; return to the study unit for specified study visits; and able to participate in the study for the entire period.
3. Patient is classified as New York Heart Association/World Health Organisation (NYHA/WHO) functional Class I, II or III.
4. Patient has CardioMEMS PA Sensor implanted and has completed treatment per parent protocol in Phase 2 Study CS1-003.
5. Female patient of childbearing potential must be willing and able to practice effective contraception during the study and continuing contraception for 30 days after their last dose of study drug. A female patient of non-childbearing potential is defined as being surgically sterilized by bilateral tubal ligation, bilateral oophorectomy, or hysterectomy. A female patient 45 to 60 years of age, who is post-menopausal for at least 1 year, and has a follicle-stimulating hormone level confirmation indicating post menopausal status will be considered of non-childbearing potential. A female patient >60 years of age is considered post menopausal and of non childbearing potential.

Exclusion Criteria:

1. Patient has a concomitant medical disorder that is expected to limit the patient's life-expectancy to ≤1 year.
2. Patient has thrombocytopenia: platelets <100,000/mm3.
3. Patient has a recent history of pancreatic disease.
4. Patient is a pregnant or lactating female.
5. Patient has active coronavirus disease 19 (COVID-19); however, those with previous COVID 19 are permitted.
6. Patient is participating in another investigational study which, in the opinion of the Investigator, would interfere with the study compliance or outcome assessments.
7. Patient is on regular treatment with other anti-epilepsy drugs or other prohibited medications (See Section 6.8.1) that cannot be discontinued at Roll-over or Restart Visit (V1).
8. Patient is on regular anticoagulation or on antiplatelet therapy that cannot be discontinued. A low daily dose aspirin (<125 mg) is allowed, ie, "baby" aspirin.
9. Patient has significant liver dysfunction as measured by any one of the following at Roll-over or Restart Visit (V1) (including patients with acute or chronic hepatitis as well as patients with own or family history of serious hepatitis, especially drug related):

   1. Alanine aminotransferase (ALT) >2.0 × upper limit of normal (ULN).
   2. Aspartate aminotransferase (AST) >2.0 × ULN.
   3. Serum bilirubin ≥1.6 mg/dL or >2.0 × ULN.
10. Patient with any major surgical procedure or trauma within 30 days prior to Roll-over or Restart Visit (V1) or planned surgical procedure during the study period.
11. Patient has known hypersensitivity to study drug or any of the excipients of the drug formulation.
12. Patient prematurely discontinued CS1 treatment in parent Study CS1-003 due to safety concerns of the Investigator.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Fredrik Frick, Gothenburg, Sweden